CLINICAL TRIAL: NCT05573178
Title: Different Catheter Ablation Strategy in Vasovagal Syncope: A Single Center, Prospective, Randomized Study
Brief Title: Different Catheter Ablation Strategy in Vasovagal Syncope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Yan Yao, MD,PhD, Chief of First Department of Arrythmia Center, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019XK320059
Record Dates: First submitted 2021-01-27; First posted 2022-10-10 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Syncope, Vasovagal
Keywords: Vasovagal syncope; cardioneuroablation
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ablation of left atrial ganglion plexus (Experimental): In this arm, ablation of GPs will only performed in the left atrium, including ablation of right anterior ganglion plexus (RAGP)，left superior ganglion plexus (LSGP)，left ganglion plexus (LLGP), left interior ganglion plexus (LIGP) and right interior ganglion plexus（RIGP).
  Interventions: Procedure: cardiac ganglion plexus ablation(cardioneuroablation)
- combined ablation of left and right atrial ganglion plexus (Experimental): In the arm the, ablation of GPs will perform in both atrium, including ablation of right anterior ganglion plexus (RAGP)，left superior ganglion plexus (LSGP)，left ganglion plexus (LLGP), left interior ganglion plexus (LIGP), right interior ganglion plexus (RIGP), and superior vena cava ganglion plexus (SVCGP). SVCGP were ablated in the right atrium，the left GPs were ablated through the left atrium
  Interventions: Procedure: cardiac ganglion plexus ablation(cardioneuroablation)

INTERVENTIONS:
Procedure: cardiac ganglion plexus ablation(cardioneuroablation) — Under the guidance of three-dimensional system, the located ganglion plexus was ablated with saline irrigating electrode. The upper limit of power was 40W, the upper limit of temperature was 43 ℃, and the washing rate of saline was 17ml/min. The site of vagal reaction during ablation was defined as the effective ablation site. The surgical end point of denervated interventional therapy is defined as the disappearance of vagal response at the effective ablation site or the ablation of each effective point discharge for at least 30 seconds.

SUMMARY:
This study is a prospective, single-center randomized controlled clinical trial. patients with refractory vasovagal syncope were randomly divided into two groups according to the proportion of 1:1. Group A: simple left atrial ganglion plexus ablation (RAGP + LSGP + LLGP + LIGP + RIGP ablation); B group: left atrial ganglion plexus combined with right atrial ganglion plexus ablation (group A + consolidation ablation of RAGP at the junction of right atrial septum and superior vena cava). To clarify the role of RAGP in cardiac autonomic nervous system and the effect of ablation, to establish the standard stragtegy of cardiac nerve ablation.

DETAILED DESCRIPTION:
Vasovagal syncope (VVS) is the most common syncope type in clinic, but routine therapy shows no benefits. Cardiac nerve ablation affects the function of cardiovascular system by accurately mapping and ablation of cardiac autonomic ganglion plexus and adjusting cardiac sympathetic-vagal balance. The existing clinical evidence is mostly exploratory or registered clinical studies, and the sample size is small. This study intends to adopt a prospective, randomized controlled study to compare the efficacy of simple left atrial ganglion plexus ablation and left atrial ganglion plexus ablation combined with right atrial ganglion plexus ablation in the treatment of VVS, and to establish the relevant cardiac nerve ablation standards.

This study is a prospective, single-center randomized controlled clinical trial. patients with refractory vasovagal syncope were randomly divided into two groups according to the proportion of 1:1. Group A: simple left atrial ganglion plexus ablation (RAGP + LSGP + LLGP + LIGP + RIGP ablation); B group: left atrial ganglion plexus combined with right atrial ganglion plexus ablation (group A + consolidation ablation of RAGP at the junction of right atrial septum and superior vena cava).

Atrial modeling was established under the guidance of Ensite three-dimensional mapping system, and then MicroPace EPS 320 was used to stimulate and induce the main distribution areas of autonomic ganglia. The high frequency stimulation mode is set as follows: the stimulation frequency is 20 Hz, the voltage is 10 to 20 volts, and the pulse width is 5 milliseconds. The main sites of high frequency stimulation include: the left superior pulmonary vein and the left atrial posterior wall of LSGP, the left inferior pulmonary vein orifice of LIGP, the LLGP, around the right inferior pulmonary vein orifice, the RIGP, around the right superior pulmonary vein and the left atrial junction of the right superior pulmonary vein, the right atrial septum of RAGP, and the superior vena cava junction to stimulate RAGP. Ganglion localization standard: locate the site of vagal response (ventricular arrest, atrioventricular block, RR interval prolongation at least 50%) after high frequency stimulation, and mark it in the three-dimensional model.

Under the guidance of three-dimensional system, the located ganglion plexus was ablated with saline irrigating electrode. The upper limit of power was 40W, the upper limit of temperature was 43 ℃, and the washing rate of saline was 17ml/min. The site of vagal reaction during ablation was defined as the effective ablation site . Denervated interventional therapy. The surgical end point of the treatment was defined as the disappearance of vagal response at the effective ablation site or the ablation of each effective point discharge for at least 30 seconds. Cardiac electrophysiological parameters such as heart rate, AH interval, HV interval, recovery time of sinoatrial node, Wenckebach point of atrioventricular conduction and atrioventricular conduction refractory period were measured before and after ablation.

The patients were followed up at 3 months, 6 months, 12 months and 24 months respectively after ablation procedure, to observe whether there were recurrent syncope and /or pre-syncope (including the time and frequency of recurrent syncope, inducing factors, and whether complicated with fall injury, etc.), and to reassessed tilt test, 24-hour ambulatory electrocardiogram and fill in Short Form-36 (SF-36) and Euroqol (EQ-5D) quality of life score form. To evaluate the safety and efficacy of cardiac nerve ablation in the prevention of refractory vasovagal syncope. The tilt test, the changes of vagus nerve function and the improvement of quality of life before and after were analyzed and compared. To evaluate the efficacy and safety of cardiac nerve ablation strategies, and to explore the role and optimization of RAGP in cardiac nerve ablation.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form.
* Definitely diagnosed as vasovagal syncope (according to the 2018 ESC syncope diagnosis and management guidelines).
* Positive head-up tilt test (cardiac inhibition type, mixed type).
* Syncope attacks ≥ 3 times in 1 year before operation and/or recurrence of syncope in the last 6 months.
* More than 2 kinds of routine treatment were ineffective or could not tolerate their side effects.

Exclusion Criteria:

* Syncope caused by other causes.
* Heart failure (NYHA grade Ⅲ or IV), congenital heart disease, valvular heart disease, deficiency. Bloody heart disease, hypertrophic cardiomyopathy, dilated cardiomyopathy, arrhythmogenic cardiomyopathy and myocarditis, chronic. Hepatic and renal insufficiency, diabetes, nervous system diseases, etc.
* Acute coronary syndrome or myocardial infarction occurred in recent 6 months; cerebrovascular events occurred in recent 3 months (such as short. Transient ischemic attack, stroke) or other disturbance of cerebral blood supply.
* Previously undergone cardiac catheter ablation, cardiac surgery and / or permanent cardiac pacemaker implantation.
* Left atrial thrombus and / or left atrial diameter > 55mm or EF < 35% were found by echocardiography or CT.
* Pregnancy and lactation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with syncope during follow up | 12 month after ablation procedure
  Syncope was defined as a transient loss of consciousness and complete recovery in a very short time. We documented each time that syncope occurred.
Number of Participants with pre-syncope during follow up | 12 month after ablation procedure
  Pre-syncope was defined as the prodrome before syncope, such as dizziness, sweating， dyspnea, and paleness, and patients did not actually fall down. We documented each time that syncope occurred.

SECONDARY OUTCOMES:
Number of Participants with positive results of head-upright tilt test | 6 month after ablation procedure
  the positive results of head-upright tilt test were defined by VASIS standard
Number of Participants with positive results of head-upright tilt test | 12 month after ablation procedure
  the positive results of head-upright tilt test were defined by VASIS standard
changes of deceleration capacity compare to baseline | 3 days after ablation procedure
  The deceleration capacity was calculated with the 24-hour ambulatory electrocardiogram through the phase-rectified signal averaging technique.
changes of deceleration capacity compare to baseline | 3 month after ablation procedure
  The deceleration capacity was calculated with the 24-hour ambulatory electrocardiogram through the phase-rectified signal averaging technique.
changes of deceleration capacity compare to baseline | 6 month after ablation procedure
  The deceleration capacity was calculated with the 24-hour ambulatory electrocardiogram through the phase-rectified signal averaging technique.
changes of deceleration capacity compare to baseline | 9 month after ablation procedure
  The deceleration capacity was calculated with the 24-hour ambulatory electrocardiogram through the phase-rectified signal averaging technique.

CONTACTS AND LOCATIONS:
Overall Officials: Yao yan, PhD, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases
Locations (2):
- China (2):
  - China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality
  - Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hu F, Zheng L, Liu S, Shen L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Avoidance of Vagal Response During Circumferential Pulmonary Vein Isolation: Effect of Initiating Isolation From Right Anterior Ganglionated Plexi. Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007811. doi: 10.1161/CIRCEP.119.007811. Epub 2019 Nov 25. PMID 31760820
- [Result] Zhu C, Hanna P, Rajendran PS, Shivkumar K. Neuromodulation for Ventricular Tachycardia and Atrial Fibrillation: A Clinical Scenario-Based Review. JACC Clin Electrophysiol. 2019 Aug;5(8):881-896. doi: 10.1016/j.jacep.2019.06.009. Epub 2019 Aug 19. PMID 31439288
- [Derived] Tu B, Chen A, Cai S, Zhang Z, Zhou L, Lai Z, Maimaitijiang P, Hu Z, Wu L, Ding L, Zheng L, Yao Y. The Efficacy of Left Atrial vs Biatrial Cardioneuroablation in Patients With Vasovagal Syncope: A Randomized Clinical Trial. JACC Clin Electrophysiol. 2025 Jun;11(6):1265-1276. doi: 10.1016/j.jacep.2025.01.019. Epub 2025 Mar 19. PMID 40117421
- See also: article on pubmed — http://pubmed.ncbi.nlm.nih.gov/31760820/
- See also: article on pubmed — http://pubmed.ncbi.nlm.nih.gov/31439288/